CLINICAL TRIAL: NCT03465995
Title: Test and Evaluation of Non-Invasive Neuro-Assessment Devices (NINAD: Neurokinetics, Inc, iPAS
Acronym: NINADiPAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: The Citadel, The Military College of North Carolina (Unknown)
Responsible Party: Sponsor
Other Study IDs: MEM 91-2714
Record Dates: First submitted 2017-06-20; First posted 2018-03-15 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Traumatic Brain Injury; Post Traumatic Stress Disorder
MeSH Terms: conditions — Brain Injuries, Traumatic; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- NKI iPAS Diagnostic Protocol: Research participants who qualify for this study will put on EKG leads, and then a non-invasive device called iPAS, which will record heart rate and eye tracking data while participants perform a task on the screen of the device. The testing session will not exceed 30 minutes. Participants will take a total of 3 recordings over a period of roughly 5 weeks.
  Interventions: Device: NKI i-PAS Diagnostic Protocol

INTERVENTIONS:
Device: NKI i-PAS Diagnostic Protocol — The NKI i-PAS:
  The NeuroKinetics i-PAS system is a mobile assessment device with an integrated display for eye tracking with the following properties: a head mounted display, a sampling rate of 100 frames per second, eye tracking in the horizontal, vertical and torsional axes, and pupil area measurement with a spatial resolution less than 0.1 o. The testing protocol includes: optokinetic tracking, smooth pursuit horizontal, smooth pursuit vertical, saccade random horizontal, saccade random vertical, saccade predictive horizontal, antisaccade (horizontal), self-paced saccade, saccade and reaction times, visual reaction time, auditory reaction time, gaze horizontal, light reflex, subjective visual (vertical) and subjective vertical horizontal. Several quantitative measures are computed from the data acquired in each test, and these measures are then employed in a multivariate diagnostic assessment.

SUMMARY:
The long term goal for the Traumatic Injury Research Program (TIRP) is testing of novel devices for the identification and longitudinal assessment of traumatic brain injury (TBI). DoD (United States Department of Defense) has now tasked TIRP with the test and evaluation of these devices to assess reliability and validity. The objective of this effort is to test the reliability of the NKI, Inc, (NeuroKinetics, Inc) i-PAS device using a test/re-test protocol with healthy controls.

The research design is test/re-test, with three assessments obtained on three separate visits. This will allow the assessment of reliability of both the device and the measure(s) that are computed from the input signals. Participants will be Healthy Controls (HC) as defined in the inclusion exclusion section.

In this initial study, investigators will be administering standardized self-report instruments (Standard Form 36 - SF36, and Symptom Checklist 90r, or SCL-90r), standard three-lead EKG. In addition they will administer the NKI i-PAS specific protocol as delineated by NKI.

DETAILED DESCRIPTION:
Traumatic brain injury is not only a significant medical and operational issue for the military but is a significant public health issue in the United States. The CDC reports that 1.4 million Americans sustain traumatic brain injuries each year. Of these 50,000 die, 235,000 are hospitalized and 1.1 million are treated and released from the emergency department. Among children fourteen years old and younger, there are an estimated 2685 TBI deaths per year, 37,000 hospitalizations and 435,000 emergency room visits.

Additionally, the Centers for Disease Control (CDC) also notes that TBI is significantly under-reported.

Traumatic brain injury is under detected. Neuropsychological evaluations are often nondisclosing The DoD has invested considerable funds in the development of devices for use in acute and chronic assessment of TBI. Unfortunately none of these devices have been tested systematically to establish reliability of the equipment, reliability of the signals obtained, or reliability of the measures derived from the signals obtained.

The NeuroKinetics i-PAS system is a mobile assessment device with an integrated display for eye tracking with the following properties: a head mounted display, a sampling rate of 100 frames per second, eye tracking in the horizontal, vertical and torsional axes, and pupil area measurement with a spatial resolution less than 0.1 o. The testing protocol includes: optokinetic tracking, smooth pursuit horizontal, smooth pursuit vertical, saccade random horizontal, saccade random vertical, saccade predictive horizontal, antisaccade (horizontal), self-paced saccade, saccade and reaction times, visual reaction time, auditory reaction time, gaze horizontal, light reflex, subjective visual (vertical) and subjective vertical horizontal. Several quantitative measures are computed from the data acquired in each test, and these measures are then employed in a multivariate diagnostic assessment.

It is important to distinguish between a device, a signal and a measure. As used here, the term device refers to a hardware technology used to obtain a signal. In the case of neurodiagnostic devices, the signal is usually a measurement of voltage as a function of time. Examples of signals pertinent to the present discussion include the electrocardiogram (providing an assessment of autonomic nervous system status), the electroencephalogram, evoked potentials, event related potentials, balance records and eye movement trajectories. A clear distinction must be drawn between a signal, typically a voltage record, and a measure which is a number that is computed from the voltage signal. Reliability and validity must be investigated separately for each measure For example, a dozen measures may be calculated from the same EEG voltage signal. The reliability and validity of each measure must be evaluated.

The objectives of this initial study are limited. The investigators address the question: are the measures obtained from the NeuroKinetics iPAS eye tracking system longitudinally stable in a clinically stable healthy participant? These measures are described in a subsequent section.

A single channel ECG will be acquired and measures of heart rate variability will be calculated from this signal. Measures of heart rate variability provide an indirect surrogate measure of complex multifactorial states that can have an impact on psychophysiological variables. Alterations of heart rate variability (HRV) are associated with pain, attention and cognitive function and fatigue, all of which can affect neurophysiological measures. High intra-individual variability in a test-retest study is a warning sign that between recording changes in the state of the participant rather than reliability failures in the eye tracking measure may be playing a role in low reliability.

Following consent, eligibility will be established based on head injury history, the score on the Symptom Checklist 90 (in the Supporting Documents file), the Short Form 36 (in the Supporting Documents file), and the Defense Veterans Brain Injury Center (DVBIC) Three Question Screening Tool.

The standard iPAS eye tracking evaluation as described below will be administered and the ECG will be recorded simultaneously during this process.

A second recording will be obtained within two to six days of the first recording.

A third recording will be obtained at approximately four weeks following the first recording.

This study will establish normal values of neuroassessment measures obtained from healthy controls and will be used to establish the statistical separation between healthy populations and clinical populations presenting neuropsychiatric disorders including TBI-positive patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants
* Between 18 and 55 years old
* In good general health. Good general health is operationalized for the purpose of this study by scores within one standard deviation of the mean in all eight sections of the short form 36.
* A normalized Global Severity Scale of less than or equal to 65 on the Symptom Checklist 90-R and subscale scores less than the cut scores indicating significant pathology.

Exclusion Criteria:

* Traumatic brain injury positive as determined by the DVBIC 3 Question Screening Tool.
* Any history of seizures or Central Nervous System (CNS) tumors
* A normalized Global Severity Scale of more than 65 on the Symptom Checklist 90-R or any subscale score indicating significant pathology.
* Scores greater than one standard deviation from the mean on all eight sections of the Short Form 36.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Students of the The Citadel, South Carolina.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-02-22 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Unit performance reliability | Total participant time burden for the study is roughly 2 hours over the course of 5 weeks.
  Due to the non-interventional nature of this study, no outcome data will be collected or tracked. A database of baseline performance profiles will be developed for a group of healthy research participants. The ultimate outcome of this study is a determination of reliability for the device.

CONTACTS AND LOCATIONS:
Locations (1):
- The Citadel, Charleston, South Carolina, United States